CLINICAL TRIAL: NCT03726658
Title: A Two-Part, Double-Blind, Placebo-Controlled, Single- and Multiple-Dose (Part A) or Twice Daily Dose (Part B) Study of AGN-241751 in Adult Participants With Major Depressive Disorder
Brief Title: AGN-241751 in the Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Syndeio Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3125-104-002
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AGN-241751 3mg (Experimental): AGN-241751, oral administration, once per day in Part A. Twice per day (BID) in Part B
  Interventions: Drug: AGN-241751
- AGN-241751 10mg (Experimental): AGN-241751, oral administration, once per day
  Interventions: Drug: AGN-241751
- AGN-241751 25mg (Experimental): AGN-241751, oral administration, once per day in Part A. Twice per day (BID) in Part B
  Interventions: Drug: AGN-241751
- Placebo (Placebo Comparator): Placebo, oral administration, once per day in part A. Twice per day (BID) in Part B
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGN-241751 — AGN-241751 is supplied in tablet form
  Arms: AGN-241751 10mg; AGN-241751 25mg; AGN-241751 3mg
Drug: Placebo — Placebo is supplied in tablet form
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of AGN-241751 in participants with Major Depressive Disorder

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the participant has been obtained prior to any study-related procedures
* Meet DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) criteria (American Psychiatric Association, 2013). for MDD (based on confirmation from the modified SCID), with a current major depressive episode of at least 8 weeks and not exceeding 18 months in duration at Visit 1.
* Have a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test at screening (Visit 1) if a WOCBP (Women of Childbearing Potential).
* Female participants willing to minimize the risk of becoming pregnancy for the duration of the clinical study and follow-up period. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
* Not a WOCBP (Women of Childbearing Potential). OR
* A WOCBP (Women of Childbearing Potential). who agrees to follow the contraceptive guidance in during the treatment period and for at least 4 to 5 weeks after the last dose of study treatment.
* Male participants willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period. A male participant must agree to use contraception during the treatment period and for at least 10 weeks after the last dose of study treatment and refrain from donating sperm during this period.
* Able, as assessed by the investigator, and willing to follow study instructions and likely to complete all required study visits.

Exclusion Criteria:

Psychiatric and Treatment-Related Criteria

* DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) based diagnosis of any disorder other than MDD that was the primary focus of treatment within 6 months before Visit 1. Comorbid generalized anxiety disorder, social anxiety disorder, or specific phobias are acceptable provided they play a secondary role in the balance of symptoms and are not the primary driver of treatment decisions.
* Lifetime history of meeting DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition)criteria for:
* Schizophrenia spectrum or other psychotic disorder
* Bipolar or related disorder
* Major neurocognitive disorder
* Neurodevelopmental disorder of greater than mild severity or of a severity that impacts the participant's ability to consent, follow study directions, or otherwise safely participate in the study
* Dissociative disorder
* Posttraumatic stress disorder
* MDD with psychotic features
* History of meeting DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, 5th Edition) criteria for alcohol or substance use disorder (other than nicotine or caffeine) within the 6 months before Screening (Visit 1).
* History (based on participant report and/or medical records, and investigator judgment) of the following:
* Inadequate response to ECT, a monoamine oxidase inhibitor, ketamine, or adjunctive treatment with an antipsychotic
* Treatment with clozapine or any depot antipsychotic
* ECT, vagus nerve stimulation, transcranial magnetic stimulation, or any experimental central nervous system treatment during the current episode or in the 6 months before Screening (Visit 1) whichever is longer)
* Tardive dyskinesia, serotonin syndrome, or neuroleptic malignant syndrome
* Having received:
* Anticonvulsant/mood stabilizer, within 1 year prior to Screening (Visit 1)
* Antipsychotic in the current episode, with the exception of quetiapine given for insomnia ≤ 50 mg/day provided it can be safely discontinued prior to Visit 2
* Combination therapy of more than 2 ADTs in the current episode if given for depression at adequate dose and duration
* ADT augmentation agent in the current episode
* Lifetime history of nonresponse to ≥ 2 antidepressants after adequate trials (adequate treatment is defined as at least 6 weeks at an adequate dose(s) based on approved package insert recommendations).
* Positive result at Screening (Visit 1) from the UDS (Urine Drug Screen) test for any prohibited medication. Exception: Participants with a positive UDS (Urine Drug Screen) at Screening for opiates, cannabinoids, or episodic use of benzodiazepines may be allowed in the study provided:
* The drug was used for a legitimate medical purpose;
* The drug can be safely discontinued prior to participation in the study (except for episodic use of benzodiazepines which may be continued); and
* A repeat UDS is negative for these substances prior to enrollment (except for episodic use of benzodiazepines which may be continued)
* Part B participants who have regularly been using benzodiazepines (even for legitimate medical purposes) for more than 2 months should not be included in the study if there is doubt that the medication can be safely discontinued during screening.
* A suicide attempt within the past year
* Prior participation in any investigational study of AGN-241751
* Initiation or termination of psychotherapy for depression within the 3 months preceding Screening (Visit 1), or plans to initiate, terminate, or change such therapy during the course of the study. (Support meetings or counseling [eg, marital counseling] are allowed provided they are no more frequent than weekly and do not have treatment of depression as their objective.)
* Ongoing treatment with phototherapy, or termination of phototherapy within 1 month of Visit 1.
* Known allergy or sensitivity to the study medication or its components.
* Hypothyroidism or hyperthyroidism, unless stabilized on appropriate pharmacotherapy with no change in dosage for at least 1 month before Screening (Visit 1)
* History of seizure disorder, stroke, significant head injury, tumor of the central nervous system, or any other condition that predisposes to seizure.
* Known HIV infection
* Part B: Previously diagnosed hearing loss; current hearing aid users (within the last 6 months), or history of gross hearing loss, such as conductive hearing loss, congenital hearing loss, sudden hearing loss, hearing loss due to recent noise or occupational exposure.
* Current enrollment in an investigational drug or device study or participation in such a study within 6 months of entry into this study (or within 3 months of entry into this study (Part B).
* Part B: Prior participation in any investigational study of AGN-241751, rapastinel, ketamine, or esketamine. Part B participants should not have participated in Part A at any time, and Part A participants should not have participated in Part B at any time (ie, Part A is not a contingent step to participate in Part B).
* Employee, or immediate relative of an employee, of the sponsor, any of its affiliates or partners, or the study center
* Inability to speak, read, and understand the English language sufficiently to understand the nature of the study, to provide written informed consent, or to allow the completion of all study assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2019-10-23 (Actual); Study Completion 2019-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M Burch, MD PhD, Study Director — Syndeio Biosciences, Inc
Locations (5):
- United States (5):
  - Alea Research, Phoenix, Arizona
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Hassman Research Institute, Berlin, New Jersey
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AGN-241751 3mg Daily; AGN-241751 10mg Daily; AGN-241751 25mg Daily: AGN-241751, oral administration, once per day in Part A.
  AGN-241751: AGN-241751 is supplied in tablet form
- Placebo Daily: Placebo, oral administration, once per day in part A.
  Placebo: Placebo is supplied in tablet form
- AGN-241751 3mg Two Times Per Day; AGN-241751 25mg Two Times Per Day: AGN-241751, oral administration, BID in Part B.
  AGN-241751: AGN-241751 is supplied in tablet form
- Placebo 2 Times Per Day: Placebo, oral administration, two times per day in part B.
  Placebo: Placebo is supplied in tablet form
Period: Overall Study
Arm/Group | AGN-241751 3mg Daily | AGN-241751 10mg Daily | AGN-241751 25mg Daily | Placebo Daily | AGN-241751 3mg Two Times Per Day | AGN-241751 25mg Two Times Per Day | Placebo 2 Times Per Day
Started | 26 | 26 | 26 | 25 | 40 | 40 | 41
Completed | 25 | 26 | 24 | 25 | 34 | 35 | 36
Not Completed | 1 | 0 | 2 | 0 | 6 | 5 | 5
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 6 | 4 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants in Part A and Part B were analyzed completely separately.
Groups:
- Total: Total of all reporting groups
Arm/Group | AGN-241751 3mg Daily | AGN-241751 10mg Daily | AGN-241751 25mg Daily | Placebo Daily | AGN-241751 3mg Two Times Per Day | AGN-241751 25mg Two Times Per Day | Placebo 2 Times Per Day | Total
Number analyzed (Participants) | 26 | 26 | 26 | 25 | 40 | 40 | 41 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (13.14) | 39.0 (13.84) | 41.4 (15.03) | 36.2 (12.43) | 38.5 (12.62) | 40.3 (14.21) | 37.7 (14.06) | 40.2 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Part A: Female | 18 | 16 | 18 | 14 | 20 | 14 | 12 | 112
  Part A: Male | 8 | 10 | 8 | 11 | 20 | 26 | 29 | 112
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 14 | 18 | 15 | 12 | 16 | 12 | 103
  Black | 9 | 11 | 7 | 8 | 25 | 22 | 26 | 108
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 5
  American Indian or Alaska Native | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 3
  Native Hawaiian or Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Multiple | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 4
  Missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 26 | 25 | 40 | 40 | 41 | 224
Montgomery-Asberg Depression Severity (MADRS) score at baseline (prior to first dose) [Mean (Standard Deviation); unit: units on a scale] — Efficacy will be measured by improvement in Montgomery-Asberg Depression Rating Scale (MADRS) total score. The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. The MADRS score ranges from 0 to 60 with a higher score indicating greater depression. A negative change score indicates improvement. Results are reported as change from baseline in treated group compared to change from baseline in placebo, reported as least squares difference and (standard error) calculated from a mixed model-repeated measures analysis
  units on a scale | 34.0 (4.48) | 35.0 (4.51) | 33.3 (5.02) | 34.0 (4.20) | 34.1 (3.62) | 34.2 (4.12) | 33.8 (5.05) | 34.06 (0.509)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change in MADRS Score at 1 Day the Initial Dose of AGN-241751 Reported as Change From Baseline in Treated Group Compared With Change From Baseline in Placebo Group
Description: Efficacy will be measured by improvement in Montgomery-Asberg Depression Rating Scale (MADRS) total score. The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. The MADRS score ranges from 0 to 60 with a higher score indicating greater depression. A negative change score indicates improvement. Results are reported as change from baseline in treated group compared to change from baseline in placebo, reported as least squares difference and (standard error) calculated from a mixed model-repeated measures analysis
Time Frame: Baseline (Day1) to Day 2
Population: Modified Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AGN-241751 3mg Daily | AGN-241751 10mg Daily | AGN-241751 25mg Daily | Placebo Daily | AGN-241751 3mg Two Times Per Day | AGN-241751 25mg Two Times Per Day | Placebo 2 Times Per Day
Number analyzed (Participants) | 26 | 26 | 26 | 25 | 0 | 0 | 0
score on a scale | -9.4 (1.57) | -6.7 (1.58) | -9.5 (1.57) | -9.3 (1.61) |  |  |
Statistical Analysis 1: Comparison: AGN-241751 3mg Daily vs Placebo Daily; Change from baseline in treated group compared to change from baseline in placebo group on Day 2 (Day 1 post initial dose). Since this was a phase 1 study no power calculation was performed; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 2 (Day 1 post initial dose). Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; p = 0.98, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -0.1, Standard Error of Mean 2.24
Statistical Analysis 2: Comparison: AGN-241751 10mg Daily vs Placebo Daily; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.25, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Change from baseline in treated group compared to change from baseline in placebo group on Day 2 (Day 1 post initial dose); Median Difference (Final Values) = 2.6, Standard Error of Mean 2.25
Statistical Analysis 3: Comparison: AGN-241751 25mg Daily vs Placebo Daily; Change from baseline in treated group compared to change from baseline in placebo group on Day 2 (Day 1 post initial dose); Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 2 (Day 1 post initial dose); p = 0.93, Mixed Models Analysis — Change from baseline in treated group compared to change from baseline in placebo group on Day 2 (Day 1 post initial dose); Mean Difference (Final Values) = -0.2, Standard Error of Mean 2.26

2. Primary Outcome: Part B: Change From Baseline in MADRS Score at Day 8 Post the Initial Dose of AGN-241751 (i.e. 1 Day After the Seventh Daily Dose)
Description: Efficacy was measured by improvement in Montgomery-Asberg Depression Rating Scale (MADRS) total score. The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. The MADRS score ranges from 0 to 60 with a higher score indicating greater depression. A negative change score indicates improvement.
Time Frame: Baseline (Day 1) to Day 8
Population: Modified Intent-to-Treat, subjects who completed Day 8 assessments
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AGN-241751 3mg Daily | AGN-241751 10mg Daily | AGN-241751 25mg Daily | Placebo Daily | AGN-241751 3mg Two Times Per Day | AGN-241751 25mg Two Times Per Day | Placebo 2 Times Per Day
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 37 | 38 | 40
score on a scale |  |  |  |  | -12.8 (1.53) | -10.5 (1.52) | -10.9 (1.48)
Statistical Analysis 1: Comparison: AGN-241751 3mg Two Times Per Day vs Placebo 2 Times Per Day; Chane from baseline in treated group compared to change from baseline in placebo group. Since this was a phase 1 study no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group; p = 0.43, Mixed Models Analysis — a priori threshold for statistical significance was <0.05; Mean Difference (Final Values) = -1.6, Standard Error of Mean 2.02
Statistical Analysis 2: Comparison: AGN-241751 25mg Two Times Per Day vs Placebo 2 Times Per Day; Change from baseline in treated group compared to change in placebo group. Since this was a phase 1 study no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change in baseline in placebo group; p = 0.84, Mixed Models Analysis — The a priori threshold for statistical significance was P <0.05; Median Difference (Final Values) = 0.4, Standard Error of Mean 2.02

3. Secondary Outcome: Part A: Change From Baseline in MADRS Score on Day 9 and Day 15 of AGN-241751 Once Daily and at Day 22 (7 Days After Completion of AGN-241751 Dosing) Compared With Change in Placebo
Description: as for outcome 2
Time Frame: Baseline (Day 1) to Day 22
Population: Modified Intent-to-Treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AGN-241751 3mg Daily | AGN-241751 10mg Daily | AGN-241751 25mg Daily | Placebo Daily | AGN-241751 3mg Two Times Per Day | AGN-241751 25mg Two Times Per Day | Placebo 2 Times Per Day
Number analyzed (Participants) | 26 | 26 | 26 | 25 | 0 | 0 | 0
score on a scale
  Day 9 | -13.0 (1.86) | -13.6 (1.87) | -14.1 (1.85) | -12.0 (1.89) |  |  |
  Day 15: number analyzed (Participants) | 26 | 26 | 24 | 25 | 0 | 0 | 0
  Day 15 | -13.2 (1.86) | -13.7 (1.87) | -13.2 (1.89) | -11.6 (1.90) |  |  |
  Day 22: number analyzed (Participants) | 23 | 25 | 26 | 23 | 0 | 0 | 0
  Day 22 | -12.5 (1.97) | -11.8 (1.91) | -14.5 (1.90) | -13.6 (1.94) |  |  |
Statistical Analysis 1: Comparison: AGN-241751 3mg Daily vs Placebo Daily; Change in MADRS score in treated groups compared to placebo group on Day 9. Since this was a phase 1 study no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 9; p = 0.69, Mixed Models Analysis — A priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -1.1, Standard Error of Mean 2.65
Statistical Analysis 2: Comparison: AGN-241751 10mg Daily vs Placebo Daily; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — Change in MADRS score in treated groups compared to placebo group on Day 9; p = 0.44, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -2.1, Standard Error of Mean 2.66
Statistical Analysis 3: Comparison: AGN-241751 25mg Daily vs Placebo Daily; [analysis description as in outcome 3, analysis 1]; Test type: Equivalence — Change in MADRS score in treated groups compared to placebo group on Day 9; p = 0.43, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = 2.1, Standard Error of Mean 2.66
Statistical Analysis 4: Comparison: AGN-241751 3mg Daily vs Placebo Daily; Change in MADRS score in treated groups compared to placebo group on Day 15. Since this was a phase 1 study no power calculaton was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change in MADRS score in treated groups compared to placebo group on Day 15; p = 0.55, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Median Difference (Final Values) = -1.1, Standard Error of Mean 2.65
Statistical Analysis 5: Comparison: AGN-241751 10mg Daily vs Placebo Daily; Change in MADRS score in treated groups compared to placebo group on Day 15. Since this was a phase 1 study no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change in MADRS score in treated groups compared to placebo group on Day 15; p = 0.44, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -2.1, Standard Error of Mean 2.66
Statistical Analysis 6: Comparison: AGN-241751 25mg Daily vs Placebo Daily; [analysis description as in outcome 3, analysis 5]; Test type: Equivalence — Change in MADRS score in treated groups compared to placebo group on Day 15; p = 0.56, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Median Difference (Final Values) = -1.6, Standard Error of Mean 2.69
Statistical Analysis 7: Comparison: AGN-241751 3mg Daily vs Placebo Daily; Change in MADRS score in treated groups compared to placebo group on Day 22. Since this was a phase 1 study no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change in MADRS score in treated groups compared to placebo group on Day 22; p = 0.80, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = 0.7, Standard Error of Mean 2.74
Statistical Analysis 8: Comparison: AGN-241751 10mg Daily vs Placebo Daily; [analysis description as in outcome 3, analysis 7]; Test type: Equivalence — Change in MADRS score in treated groups compared to placebo group on Day 22; p = 0.45, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Median Difference (Final Values) = -2.1, Standard Error of Mean 2.74
Statistical Analysis 9: Comparison: AGN-241751 25mg Daily vs Placebo Daily; [analysis description as in outcome 3, analysis 7]; Test type: Equivalence — Change in MADRS score in treated groups compared to placebo group on Day 22; p = 0.67, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -1.2, Standard Error of Mean 2.77

4. Secondary Outcome: Part B: Change From Baseline in MADRS Score on Day 11, Day 14, and Day 18 of AGN-241751 Administered Two Times Daily and on Day 21 (7 Days After Completion of Dosing) in Treated Group Compared to Change From Baseline in Placebo Group
Description: Efficacy was measured by improvement in Montgomery-Asberg Depression Rating Scale (MADRS) total score. The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. The MADRS score ranges from 0 to 60 with a higher score indicating greater depression. A negative change score indicates improvement. Results are reported as change from baseline in treated group compared to change from baseline in placebo, reported as least squares difference and (standard error) calculated from a mixed model-repeated measures analysis
Time Frame: Baseline (Day 1) to Day 21
Population: Modified Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AGN-241751 3mg Daily | AGN-241751 10mg Daily | AGN-241751 25mg Daily | Placebo Daily | AGN-241751 3mg Two Times Per Day | AGN-241751 25mg Two Times Per Day | Placebo 2 Times Per Day
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 37 | 38 | 40
score on a scale
  Day 11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 36 | 34 | 35
  Day 11 |  |  |  |  | -15.8 (1.70) | -15.2 (1.72) | -14.0 (1.67)
  Day 14: number analyzed (Participants) | 0 | 0 | 0 | 0 | 34 | 37 | 40
  Day 14 |  |  |  |  | -17.0 (1.76) | -15.3 (1.82) | -14.7 (1.71)
  Day 18: number analyzed (Participants) | 0 | 0 | 0 | 0 | 25 | 30 | 29
  Day 18 |  |  |  |  | -18.3 (1.88) | -15.0 (1.98) | -16.9 (1.86)
  Day 21 |  |  |  |  | -17.3 (1.79) | -16.5 (1.84) | -16.5 (1.74)
Statistical Analysis 1: Comparison: AGN-241751 3mg Two Times Per Day vs Placebo 2 Times Per Day; Change from baseline in treated group compared to change from baseline in placebo group on Day 11. Since this was a phase 1 study, no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 11; p = 0.43, Mixed Models Analysis — a priori threshold for statistical significance was p>0.05; Mean Difference (Final Values) = -1.9, Standard Error of Mean 2.36
Statistical Analysis 2: Comparison: AGN-241751 25mg Two Times Per Day vs Placebo 2 Times Per Day; [analysis description as in outcome 4, analysis 1]; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 11; p = 0.59, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -1.3, Standard Error of Mean 2.38
Statistical Analysis 3: Comparison: AGN-241751 3mg Two Times Per Day vs Placebo 2 Times Per Day; Change from baseline in treated group compared to change from baseline in placebo group on Day 14, Since this was a phase 1 study no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 14; p = 0.35, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -2.3, Standard Error of Mean 2.44
Statistical Analysis 4: Comparison: AGN-241751 25mg Two Times Per Day vs Placebo 2 Times Per Day; Change from baseline in treated group compared to change from baseline in placebo group on Day 14. Since this was a phase 1 study, no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 14; p = 0.82, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Mean Difference (Final Values) = -0.6, Standard Error of Mean 2.48
Statistical Analysis 5: Comparison: AGN-241751 3mg Two Times Per Day vs Placebo 2 Times Per Day; Change from baseline in treated group compared to change from baseline in placebo group on Day 18. Since this was a phase 1 study, no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 18; p = 0.61, Mixed Models Analysis; Mean Difference (Final Values) = -1.4, Standard Error of Mean 2.62
Statistical Analysis 6: Comparison: AGN-241751 25mg Two Times Per Day vs Placebo 2 Times Per Day; Change from baseline in treated group compared to change from baseline in placebo group on Day 18. Since this was a phase 1 study no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 18; p = 0.47, Mixed Models Analysis — The a priori threshold for statistical significance was P<0.05; Median Difference (Final Values) = 2.0, Standard Error of Mean 2.69
Statistical Analysis 7: Comparison: AGN-241751 3mg Two Times Per Day vs Placebo 2 Times Per Day; Change from baseline in treated group compared to change from baseline in placebo group on Day 21. Since this was a phase 1 study, no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 21; p = 0.76, Mixed Models Analysis; Mean Difference (Final Values) = -0.7, Standard Error of Mean 2.48
Statistical Analysis 8: Comparison: AGN-241751 25mg Two Times Per Day vs Placebo 2 Times Per Day; Change from baseline in treated group compared to change from baseline in placebo group on Day 21. Since this was a phase 1 study no power calculation was performed. Statistical tests were 2-sided hypothesis tests performed at the 5% level of significance; Test type: Equivalence — Change from baseline in treated group compared to change from baseline in placebo group on Day 21; p = 0.99, Mixed Models Analysis — Change from baseline in treated group compared to change from baseline in placebo group on Day 21; Median Difference (Final Values) = 0.0, Standard Error of Mean 2.51

ADVERSE EVENTS:
Time Frame: Two weeks = 14 days
Description: NOTE: All values for number of participants at risk include all participants randomized, which is greater than the number of participants who received at least one dose of drug.
Arm/Group | AGN-241751 3mg Daily | AGN-241751 10mg Daily | AGN-241751 25mg Daily | Placebo Daily | AGN-241751 3mg Two Times Per Day | AGN-241751 25mg Two Times Per Day | Placebo 2 Times Per Day
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/25 | 0/41 | 0/41 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26 | 0/25 | 0/41 | 0/41 | 1/41
Other Adverse Events (participants affected / at risk) | 6/26 | 8/26 | 6/26 | 3/25 | 15/41 | 20/41 | 22/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGN-241751 3mg Daily (N=26) | AGN-241751 10mg Daily (N=26) | AGN-241751 25mg Daily (N=26) | Placebo Daily (N=25) | AGN-241751 3mg Two Times Per Day (N=41) | AGN-241751 25mg Two Times Per Day (N=41) | Placebo 2 Times Per Day (N=41)
Abortion Induced (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — induced abortion of unwanted pregnancy
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AGN-241751 3mg Daily (N=26) | AGN-241751 10mg Daily (N=26) | AGN-241751 25mg Daily (N=26) | Placebo Daily (N=25) | AGN-241751 3mg Two Times Per Day (N=41) | AGN-241751 25mg Two Times Per Day (N=41) | Placebo 2 Times Per Day (N=41)
Headache (Nervous system disorders) | 4 (4) | 5 (5) | 4 (4) | 3 (3) | 6 (6) | 10 (10) | 14 (14)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 6 (6) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
Abnormal Dreams (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/58/NCT03726658/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT03726658/SAP_001.pdf